CLINICAL TRIAL: NCT07376044
Title: GusNIP Produce Prescription Project
Brief Title: RUSH Food is Medicine Veggie Rx - GusNIP Produce Prescription
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Traci Simmons, Director Community Health and Engagement, Rush University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23122803; 2025-70413-45380 (Other Grant/Funding Number: U.S. Department of Agriculture National Institute of Food and Agriculture)
Record Dates: First submitted 2025-12-30; First posted 2026-01-29 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Food Insecurity; Diabetes in Adults; Hypertension (HTN)
Keywords: Food Insecurity; Food is Medicine; Nutrition Security; Diet-related Chronic Disease; Produce Prescription
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Produce Prescription (Other): Receipt of fresh produce prescription boxes and produce vouchers redeemable using SNAP, alongside nutrition education and chronic disease management education.
  Interventions: Behavioral: Food is Medicine

INTERVENTIONS:
Behavioral: Food is Medicine — Fresh produce food prescription program designed to address food insecurity and increase intake of nutritious foods.

SUMMARY:
The goal of this clinical trial is to assess nutrition incentives and produce vouchers to measure the impacts of food insecurity-related chronic health conditions in adults with hypertension and/or diabetes. The main questions it aims to answer are:

* Does participation increase fruit and vegetable consumption for participants?
* Does participation reduce individual and household food insecurity?
* Does participation reduce healthcare utilization and associated costs?
* Does participation lead to improvements in diet-related health outcomes (e.g., hypertension, diabetes)?
* Does participation support the local economy by increasing participant spending at local food vendors?

Participants will:

* Receive 6 months home delivered produce prescription boxes
* Receive 6 months match of produce vouchers
* Receive nutrition education and participate in Chronic Disease Self-Management classes

DETAILED DESCRIPTION:
The clinical trial will serve up to 400 participants over the GusNIP Produce Prescription project. The primary outcome measure one is to strengthen food systems access and improve participant level dietary health quality through increased fruit and vegetable consumption; reduce overall individual and household level food insecurity; reduce healthcare use and associated costs; and support local economies through local food procurement. Rush participants with or at risk of diabetes and/or hypertension who screen positive for food insecurity and meet the requirements to participate in a Produce Prescription project are referred to the Veggie Rx program for one year participation. Vouchers for up to $40 dollars match can be used concurrently with SNAP EBT benefits at a local grocer, the project's SNAP firm partner. Data will measure improvements in fruit and vegetable consumption, food security status, diet quality, knowledge and behaviors, self-efficacy, healthcare utilization and associated costs.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years of age
* Participants receiving medical care at Rush
* Participants with a diagnosis of hypertension and/or diabetes
* Participants with a positive screen for food insecurity
* Participants eligible for medical assistance through a state plan
* Participants eligible for benefits through the SNAP program
* Participants are member of a low-income household
* Participants willing to participate for duration of the program (12-months)
* Participants residing in service area of the referring Rush clinic

Exclusion Criteria:

* Adults unable to consent
* Individuals not yet adults - infants, children, teenagers
* Incarcerated individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-02-16 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Change in Fruit and Vegetable Intake | 6 months, 12 months
  Mean change in daily servings of fruits and vegetables (FV) determined by self-reported data using 10-item Dietary Screener Questionnaire (DSQ). The 10-item DSQ scale collects intake frequency of FV including the quantity (i.e., amount) and variety (i.e., kinds) through retrospective observance of the past 30-days. Scale values range from decreased, stayed the same, increased, or does not apply, with increased FV intake correlating with improved intake, and decreased correlating with less intake. A higher score means a better outcome.
Change in Food Security Status | 6months, 12 months
  Individual and household level food security as measured using the United States Department of Agriculture 10-item United States Adult Food Security Module. Measured on a scale of severity from high to low food security, including high food security, marginal food security, low food security and very low food security with very low food security meaning a worse outcome.
Change in Healthcare Utilization and Associated Costs | 6 months, 12 months
  Changes in healthcare utilization including hospital, emergency department, and outpatient visits using Electronic Health Records and claims data.
Change in Health Outcomes Associated with Hypertension | 6 months, 12 months
  Changes in hypertension clinical biomarkers through Electronic Health Records, self-reported pre and post assessments for chronic disease self-management classes. Measured by 10 mm Hg reduction in systolic BP for participants with uncontrolled hypertension, as targeted by the intervention.
Change in Health Outcome Associated with Diabetes | 6 months, 12 months
  Changes in diabetes clinical biomarkers through Electronic Health Records, self-reported pre and post assessments for chronic disease self-management classes. Measured by changes in hemoglobin A1c (HbA1c), as targeted by the intervention.
Local Economic Support | Monthly for 1 year
  Change in participant spending through use of produce vouchers at local food vendors using Supplemental Nutrition Assistance Program/Electronic Benefits Transfer leads to local economic support. Measured by point of sale dollar value of produce voucher, dollar value of Supplemental Nutrition Assistance Program purchase (Electronic Benefits Transfer sales).

CONTACTS AND LOCATIONS:
Overall Officials: Traci Simmons, DrPHc, MPH, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
IPD may not be shared to protect participant confidentiality, and PHI. Should individual data be requested, the investigators will de-identify data. Data sharing mechanisms should be in place for inquiries regarding IPD.

REFERENCES:
- [Background] Ansell, D. A., & Lightfoot, L. E. (2021). The death gap: How inequality kills. University of Chicago Press